CLINICAL TRIAL: NCT00141024
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of the Recombinant Protein Vaccine EP-1043 and the DNA Vaccine EP HIV-1090 Given Alone or in Combination in Healthy, HIV-1-Uninfected Adult Participants
Brief Title: Safety of and Immune Response to the Experimental Preventive HIV Vaccine, EP HIV-1090, in Healthy, HIV-1 Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 064; 10059 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- 1 (Experimental): Group 1 will receive 4 vaccinations of the EP-1043 vaccine or placebo. Vaccinations will be given at Months 0, 1, 3, and 6. This group was discontinued as of 12/26/06.
  Interventions: Biological: EP HIV-1043
- 2 (Experimental): Group 2 will receive 4 vaccinations of the EP-1043 vaccine or placebo. Vaccinations will be given at Months 0, 1, 3, and 6. This group was discontinued as of 12/26/06.
  Interventions: Biological: EP HIV-1043
- 3 (Experimental): In Part B, Group 3 will receive 4 vaccinations of either the EP-1043 vaccine or placebo. Vaccinations will occur at Months 0, 1, 3, and 6. This group was discontinued as of 12/26/06.
  Interventions: Biological: EP HIV-1043
- 4 (Experimental): In Part B, Group 4 will receive 4 vaccinations of either the DNA vaccine EP-HIV-1090 or placebo. Vaccinations will occur at Months 0, 1, 3, and 6.
  Interventions: Biological: EP HIV-1090
- 5 (Experimental): In Part B, Group 5 will receive 4 vaccinations of either the protein vaccine EP-1043 plus DNA vaccine EP-HIV- 1090 or placebo. Vaccinations will occur at Months 0, 1, 3, and 6. This group was discontinued as of 12/26/06.
  Interventions: Biological: EP HIV-1043; Biological: EP HIV-1090

INTERVENTIONS:
Biological: EP HIV-1043 — Recombinant protein vaccine containing the 18 HIV proteins from HIV genes Pol, Vpu, and Gag.
  The vaccine is provided in single-use 1.1-mL vials.
  Arms: 1; 2; 3; 5
Biological: EP HIV-1090 — DNA plasmid vaccine containing the genes Gag, Pol, Vpr, Nef, Rev, and Env. The vaccine is provided in single-use 1.1-mL vials.
  Arms: 4; 5

SUMMARY:
The purpose of the study is to determine the safety of and immune response to the investigational HIV vaccine, EP HIV-1090, in HIV uninfected adults.

DETAILED DESCRIPTION:
The worldwide HIV/AIDS epidemic may only be controlled through the development of a safe and effective vaccine that will prevent HIV infection. DNA vaccines are inexpensive to construct, readily produced in large quantities, and stable for long periods of time. EP HIV-1090 is a DNA HIV CTL vaccine; the proteins for which its genes code are designed to interact with CD8 cells (CTL) and cause CD8 cell proliferation. The DNA plasmids in EP HIV-1090 code for proteins conserved among HIV subtypes A, B, C, D, F, and G, which encompass the HLA subtypes of 85% of the worldwide general population.

Participants will be enrolled in this study for 1 year. Group 4 participants will receive EP HIV-1090 or placebo at study entry and Months 1, 3, and 6. There will be 11 study visits that will occur at screening; study entry; and Months 0.5, 1, 1.5, 3, 3.5, 6, 6.5, 9, and 12. A physical exam and risk reduction/pregnancy prevention counseling will occur at each visit. Participants will be asked about their adverse experiences from vaccination at each visit. Blood and urine collection will occur at selected visits.

ELIGIBILITY:
Note: Groups 1, 2, 3, and 5 have permanently discontinued enrollment per the 12/26/06 letter of amendment.

Inclusion Criteria:

* Good general health
* Have access to a participating HIV Vaccine Trials Unit (HVTU) and are willing to be followed for the duration of the study
* Willing to receive HIV test results
* Have understanding of the study
* Willing to use acceptable forms of contraception
* Negative pregnancy test

Exclusion Criteria:

* HIV vaccines in a prior HIV vaccine trial
* Immunosuppressive medications within 168 days prior to first vaccination
* Blood products within 120 days prior to first vaccination
* Immunoglobulin within 60 days prior to first vaccination
* Live attenuated vaccines within 30 days prior to first vaccination
* Investigational research agents within 30 days prior to first vaccination
* Medically indicated subunit or killed vaccines within 14 days prior to first study vaccine administration, or allergy treatment with antigen injections within 30 days prior to first vaccination
* Current tuberculosis prophylaxis or therapy
* Clinically significant medical condition, abnormal physical exam findings, abnormal laboratory results, or past medical history that may affect current health
* Any medical, psychiatric, or social condition that would interfere with the study. More information about this criterion can be found in the protocol.
* Any job-related responsibility that would interfere with the study
* Serious adverse reaction to vaccines. A person who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Autoimmune disease or immunodeficiency
* Active syphilis infection unless the participant has completed full treatment for syphilis 6 months prior to enrollment
* Unstable asthma
* Diabetes mellitus type 1 or 2
* Thyroid disease or thyroidectomy requiring treatment
* Serious angioedema within 3 years prior to enrollment
* Uncontrolled hypertension
* Body mass index (BMI) of 40 or greater
* BMI of 35 or greater if the participant is older than 45 years, has systolic blood pressure greater than 140 mm Hg, has diastolic blood pressure greater than 90 mm Hg, smokes, or has known hyperlipidemia
* Bleeding disorder
* Malignancy unless it has been surgically removed and, in the opinion of the investigator, is not likely to recur during the study period
* Seizure disorder requiring medication within the 3 years prior to enrollment
* Absence of the spleen
* Mental illness that would interfere with the study
* Other conditions that, in the judgment of the investigator, would interfere with the study
* Pregnancy, breastfeeding, or plans to become pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by local and systemic reactogenicity signs and symptoms, laboratory measures, and adverse and serious experiences | After each injection and for 12 months following the first injection

SECONDARY OUTCOMES:
Immunogenicity as assessed by HIV-specific cellular responses assessed by interferon-gamma ELISpot assays and intracellular cytokine staining | Throughout the study
Social impacts as assessed by negative experiences or problems reported by the participants | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Xia Jin, MD, PhD, Study Chair — University of Rochester; Jorge Sanchez, MD, Study Chair — Asociación Civil Impacta Salud y Educación (IMPACTA)
Locations (3):
- United States (3):
  - San Francisco Vaccine and Prevention CRS, San Francisco, California
  - Project Brave HIV Vaccine CRS, Baltimore, Maryland
  - Univ. of Rochester HVTN CRS, Rochester, New York

REFERENCES:
- [Background] Esparza J, Osmanov S. HIV vaccines: a global perspective. Curr Mol Med. 2003 May;3(3):183-93. doi: 10.2174/1566524033479825. PMID 12699356
- [Background] Gaschen B, Taylor J, Yusim K, Foley B, Gao F, Lang D, Novitsky V, Haynes B, Hahn BH, Bhattacharya T, Korber B. Diversity considerations in HIV-1 vaccine selection. Science. 2002 Jun 28;296(5577):2354-60. doi: 10.1126/science.1070441. PMID 12089434
- [Background] Livingston BD, Newman M, Crimi C, McKinney D, Chesnut R, Sette A. Optimization of epitope processing enhances immunogenicity of multiepitope DNA vaccines. Vaccine. 2001 Sep 14;19(32):4652-60. doi: 10.1016/s0264-410x(01)00233-x. PMID 11535313
- [Background] McKinney DM, Skvoretz R, Livingston BD, Wilson CC, Anders M, Chesnut RW, Sette A, Essex M, Novitsky V, Newman MJ. Recognition of variant HIV-1 epitopes from diverse viral subtypes by vaccine-induced CTL. J Immunol. 2004 Aug 1;173(3):1941-50. doi: 10.4049/jimmunol.173.3.1941. PMID 15265928
- [Background] Wilson CC, McKinney D, Anders M, MaWhinney S, Forster J, Crimi C, Southwood S, Sette A, Chesnut R, Newman MJ, Livingston BD. Development of a DNA vaccine designed to induce cytotoxic T lymphocyte responses to multiple conserved epitopes in HIV-1. J Immunol. 2003 Nov 15;171(10):5611-23. doi: 10.4049/jimmunol.171.10.5611. PMID 14607970
- [Derived] Jin X, Morgan C, Yu X, DeRosa S, Tomaras GD, Montefiori DC, Kublin J, Corey L, Keefer MC; NIAID HIV Vaccine Trials Network. Multiple factors affect immunogenicity of DNA plasmid HIV vaccines in human clinical trials. Vaccine. 2015 May 11;33(20):2347-53. doi: 10.1016/j.vaccine.2015.03.036. Epub 2015 Mar 25. PMID 25820067